CLINICAL TRIAL: NCT06896877
Title: Assessment of the Nutritional Status and Emotional Well-being of the Worker-consumer in the Food Supply Chain.
Brief Title: Nutritional Status and Emotional Well-being of the Worker-consumer in the Food Supply Chain.
Acronym: ONEHEALTH
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Irene Giovanna Aprile, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: FDG_BRIC_ONEHEALTH
Record Dates: First submitted 2025-03-17; First posted 2025-03-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: food supply chain worker; nutritional status; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum sample will be collected from blood of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy worker: Participants will be healthy worker of the food-supply chain

SUMMARY:
The study aims to assess the well-being and safety of worker-consumers in the food industry, focusing on nutrition, musculoskeletal disorders, and regulatory policies. It follows a "OneHealth" approach, emphasizing the connection between human, animal, and environmental health. The research evaluates the nutritional status of workers in the food-supply chain, analyzing food consumption in both workplace and domestic settings to identify deficiencies or excesses. Through clinical, nutritional, and psychological assessments-including oxidative stress levels, serotonin, quality of life, and emotional well-being-the study seeks to identify high-risk groups and gender differences, providing data-driven insights for personalized dietary recommendations and targeted interventions. Findings will contribute to national policies for improved workforce well-being, supporting best practices and interventions to enhance health, safety, and productivity in the agri-food sector. The results will serve as the foundation for specific guidelines that strengthen the sector's sustainability and regulatory clarity.

DETAILED DESCRIPTION:
The study aims to assess, key health parameters in worker-consumers within the food-supply chain. The assessment will be performed during a single visit, assessing:

1. the nutritional status of workers: measuring participants' nutritional status to identify potential deficiencies or excesses.
2. biological parameters involved in stress: i) the systemic oxidative stress and serotonin levels to evaluate the potential imbalance between pro-oxidant and antioxidant; ii) the serotonin serum levels to analyze the circadian rhythm regulation and satiety perception.
3. the quality of life and emotional well-being: using online surveys and validated clinical assessment scales, the study will determine participants' quality of life, with a focus on psychological, physical, and social factors, aiming to identify potential work-related challenges in the food-supply chain.

Secondary Objectives Identification of risk groups: based on nutritional assessments and oxidative stress levels, identifying worker groups at higher risk of developing health conditions due to poor dietary habits or exposure to stress factors.

Analysis of gender differences: Investigating potential gender-based variations in nutritional status, oxidative stress levels, and quality of life, to determine whether specific dietary or health recommendations are needed for men and women.

This study is designed as an exploratory investigation aimed at comparing two groups of individuals with distinct dietary habits and lifestyle patterns, particularly focusing on sedentary workers versus non-sedentary workers engaged in physically demanding tasks.

The number of worker enrolled will be 40 (20 sedentary workers vs 20 non sedentary workers). The sample size has been determined based on existing literature evidence, utilizing phase angle (Di Vincenzo, 2011) and bioelectrical impedance vector analysis (BIVA) (Campa, 2020) as key reference parameters. Statistical power analysis was conducted using G*Power (v.3.1.9.7), employing a two-tailed independent samples t-test, with a significance level (α) set at 0.05 and 80% statistical power.

Effect size estimates (Cohen's d) were as follows: Fat Mass (FM): 0.81 (estimated power 70.1% with 20 participants per group), Fat-Free Mass (FFM): 1.30 (power >95% with 20 participants per group), BIVA Vector Length (VL): 2.06 (power 80% with only 5 participants per group). The selected sample size is sufficient to detect significant differences in FFM and VL, while for FM, the statistical power remains slightly below 80%.

ELIGIBILITY:
Inclusion Criteria:

* workers affiliated with the Experimental Center, or indirectly connected to the Experimental Center as part of the food supply chain;
* willingness to undergo specific tests, including nutritional status assessments, quality of life surveys, and emotional-affective well-being evaluations;
* signature of informed consent form.

Exclusion Criteria:

* pregnancy: pregnant women will be excluded to prevent physiological changes related to pregnancy from affecting the measurements.
* non-representative special diets: workers following special diets for medical or religious reasons, which may not be representative of the general food supply chain population, will be excluded.
* lack of signed informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy workers of food-supply-chain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
The difference in the bioimpedance vectors between two groups of patients (active workers versus sedentary workers), according to BIVA | baseline
  The difference in bioimpedance vectors between two groups of patients (active workers vs. sedentary workers) will be analyzed using Bioelectrical Impedance Vector Analysis (BIVA).
  In BIVA, the Resistance (Rz) and Reactance (Xc) of each subject, standardized by height (in meters), are plotted on an Rz-Xc graph, forming a bioimpedance vector that can be visualized and analyzed.
  Measurements will be obtained through Bioelectrical Impedance Analysis (BIA), providing raw data on Resistance (Rz) and Reactance (Xc), which reflect an individual's hydration status and body composition. The differences in bioimpedance vectors between the two groups (active vs. sedentary workers) will be assessed.

SECONDARY OUTCOMES:
Weight in kilograms | baseline
  It is a measure of body mass weight expressed in Kg
Height in meters | baseline
  It is a measure of body height expressed in meters
Body mass Index in kg/(m^2) | baseline
  It is a measure which combines the height and weight values to report Body Mass Index (BMI) expressed in kg/m²; this parameter is valid for adult men and women. World Health Organization (WHO) defined the following cut-offs for BMI corresponding to nutritional status: i. underweight <18.5; ii. normal 18.50 - 24.99; iii.overweight ≥ 25; iv. obese ≥ 30.
Waist circumferences expressed in cm | baseline
  Measures of waist circumferences expressed in cm.
Hips circumferences expressed in cm | baseline
  Measures of hips circumferences expressed in cm.
Waist-Hips Ratio (WHR) | baseline
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement (W⁄H). WHR is used as a measurement of obesity, which in turn is a possible indicator of other more serious health conditions. The WHO states that abdominal obesity is defined as a waist-hip ratio above 0.90 for males and above 0.85 for females.
Arm circumferences expressed in cm | baseline
  Measures of arm circumferences expressed in cm.
Calf circumferences expressed in cm | baseline
  Measures of calf circumferences expressed in cm.
Tissue hydration expressed in percentage from Bioelectrical Impedance Analysis (BIA). | baseline
  It provides the actual hydration values, i.e. the percentage content of fluids (Total Body Water, TBW) in the Lean Mass (Fat-Free Mass, FFM) from Bioelectrical Impedance Analysis (BIA). The values expressed in percentages (% TBW/FFM) allow immediate recognition of normo-physiological states (from 72.7 to 74.3%); any alterations towards congestion are represented with values between 74.4% - 81%, while alterations towards dehydration are identified with values between 72.6%-70%.
Nutritional index (mg 24h/height in meters) from Bioelectrical Impedance Analysis (BIA). | baseline
  Protein/energy nutrition assessment scale derived from Bioelectrical Impedance Analysis (BIA).. Creatinine excretion (Ucr/24h) is estimated by analysing the amount of cell mass detected by the sensor. The result is normalised to the subject's height and classified using the vector impedance technique into four ranges. The colour graphic representation offers simple and immediate identification of altered states of energy and/or protein malnutrition.
Resistance (Rz) from Bioelectrical Impedance Analysis (BIA). | baseline
  Resistance (Rz) is a parameter measured through Bioelectrical Impedance Analysis (BIA), reflecting the opposition of body tissues to the flow of an alternating electrical current. It is primarily influenced by the amount of total body water (TBW) and Fat-Free Mass (FFM).
Reactance (Xc) from Bioelectrical Impedance Analysis (BIA). | baseline
  Reactance (Xc) is a parameter measured through Bioelectrical Impedance Analysis (BIA), representing the capacitive properties of cell membranes and tissues. It reflects cell membrane integrity, body cell mass (BCM), and overall cellular health.
Phase Angle (PhA) from Bioelectrical Impedance Analysis (BIA). | baseline
  Phase Angle (PhA) is a parameter derived from Bioelectrical Impedance Analysis (BIA), calculated as the arctangent of reactance (Xc) to resistance (Rz). It serves as a key indicator of cell membrane integrity, cellular health, and overall nutritional status. A higher PhA is generally associated with better cellular function and nutritional status, while a lower PA may indicate malnutrition or impaired health. The phase angle expresses the proportion between intra- and extracellular spaces, describes properties about the quality of the cell and is used in the clinic as a prognostic index for chronic diseases. In a healthy adult subject, the normal value of phase angle is between 5 and 7 degrees.
Total Body Water (TBW) from Bioelectrical Impedance Analysis (BIA). | baseline
  Total Body Water (TBW) represents the total amount of water present in the body, including both intracellular water (ICW) and extracellular water (ECW). It is measured using Bioelectrical Impedance Analysis (BIA) and expressed in liters or as a percentage of body weight. TBW is a key parameter for evaluating hydration status and body composition.
Fat Free Mass (FFM) from Bioelectrical Impedance Analysis (BIA). | baseline
  Fat-Free Mass (FFM) refers to the total mass of all body components excluding fat, including muscle, bone, water, and other lean tissues. It is measured using Bioelectrical Impedance Analysis (BIA) and expressed in kilograms or as a percentage of body weight. FFM is a key indicator of muscle mass and overall body composition. Lean Mass is the compartment containing everything that is not body fat: it includes the skeleton, about 73% of body fluids, muscles, skin and organs. Good fitness assumes a FFM value of between 77-85% of body weight, depending on the subject's age.
Fat Mass (FM) from Bioelectrical Impedance Analysis (BIA). | baseline
  Fat Mass (FM) represents the total amount of body fat, measured using Bioelectrical Impedance Analysis (BIA). It is expressed in kilograms or as a percentage of body weight. FM is a key parameter for assessing body composition, nutritional status, and metabolic health. Fat Mass (FM) is a compound consisting of glycerol, a substance formed from fatty acids, which is used as an energy concentrate for the muscles. A certain amount of fat is therefore necessary both as an energy reserve and for the proper functioning of life processes. Another small amount, called essential fat, has a protective function for internal organs, but it is important that this accumulation does not exceed physiological limits. Good physical fitness presupposes a FM value of 15-23% of body weight, depending on the subject's age.
Body Cell Mass (BCM) from Bioelectrical Impedance Analysis (BIA). | baseline
  Body Cell Mass (BCM) represents the metabolically active component of Fat-Free Mass (FFM), including muscle cells, organ tissues, intracellular water, and other metabolically active cells. It is measured using Bioelectrical Impedance Analysis (BIA) and is a key indicator of nutritional status, muscle function, and overall cellular health. It is the metabolically active part of the body that does all the functional work, and the 'engine' of the body in which all major metabolic processes take place: from oxygen consumption, glucose oxidation, to protein synthesis. It is the living and active part of the organism, a compartment that the human body should be endowed with in abundance.
Skeletal Muscle Mass from Bioelectrical Impedance Analysis (BIA). | baseline
  Skeletal Muscle Mass (SMM) represents the total weight of skeletal muscles in the body, measured using Bioelectrical Impedance Analysis (BIA). It is expressed in kilograms or as a percentage of body weight and serves as a key indicator of muscle health, physical strength, and nutritional status. Skeletal Muscle Mass (SMM) accounts for about 70 % of the total muscle mass (MM).
Appendicular Skeletal Muscle Mass (ASMM) from Bioelectrical Impedance Analysis (BIA). | baseline
  Appendicular Muscle Mass (AMM) refers to the total muscle mass of the arms and legs, measured using Bioelectrical Impedance Analysis (BIA). It is expressed in kilograms or as a percentage of body weight and is a key parameter for evaluating muscle health, strength, and functional capacity. AMM is particularly relevant for assessing conditions such as sarcopenia and age-related muscle loss. It represents 75% of the Skeletal Muscle Mass (SMM) and is defined as the sum of the muscles of the upper and lower limbs. A reduction in ASMM leads to negative health consequences such as weakness, disability, a worsened quality of life.
Basal metabolic rate (BMR) from Bioelectrical Impedance Analysis (BIA). | baseline
  Basal metabolic rate (BMR) will be estimated using Bioelectrical Impedance Analysis (BIA). The estimation will be based on predictive equations integrated into the BIA device, considering factors such as fat-free mass and total body water. Basal Metabolic Rate (BMR) is the energy expenditure of an organism at rest. BMR includes the energy required for vital metabolic functions (respiration, blood circulation, digestion, nervous system activity, etc.).
Total Daily Energy Expenditure (TDEE) from Bioelectrical Impedance Analysis (BIA). | baseline
  Total Daily Energy Expenditure (TDEE) will be estimated using Bioelectrical Impedance Analysis (BIA). TDEE represents the amount of energy expended by the body at rest to sustain vital physiological functions, including circulation, respiration, and cellular metabolism. The estimation will rely on predictive equations integrated into the BIA device, providing an indirect assessment of metabolic activity, considering the basal metabolic rate (BMR) and muscular physical activity (PAL), assuming the expenditure of thermoregulation and thermogenesis as marginal.
Concentration of serum serotonin (ng/mL) | baseline
  Serum Serotonin concentration will be measured by Enzyme Linked Immunosorbent Assay (ELISA) and expressed in ng/mL
Blood concentration of haemoglobin (g/dL) | baseline
  Blood concentration of haemoglobin will be measured with colorimetric method and expressed in g/dL.
Blood levels of lymphocyte (cell per microliters or percentage) | baseline
  Lymphocyte levels in blood, expressed as absolute count (cells per microliter) or percentage of total white blood cells.
Concentration of serum albumin (g/dL) | baseline
  Serum albumin concentration will be analyzed with colorimetric method and expressed in g/dL
Concentration of serum total cholesterol (mg/dL) | baseline
  Serum concentration of total cholesterol levels measured with colorimetric method and expressed in mg/dL.
Concentration of HDL cholesterol serum levels (mg/dL) | baseline
  Serum concentration of High Density Lipoprotein (HDL) cholesterol levels measured with colorimetric method and expressed in mg/dL.
Concentration of C-reactive protein (mg/dL) | baseline
  Serum concentration of C-reactive protein levels measured with colorimetric method and expressed in mg/dL.
Concentration of glucose serum levels (mg/dL) | baseline
  Serum concentration of glucose levels measured with colorimetric method and expressed in mg/dL.
Concentration of triglycerides serum levels (mg/dL) | baseline
  Serum concentration of triglycerides levels measured with colorimetric method and expressed in mg/dL.
Concentration of magnesium serum levels (mg/dL) | baseline
  Serum concentration of magnesium levels measured with colorimetric method and expressed in mg/dL.
Concentration of calcium serum levels in mg/dL | baseline
  Serum concentration of calcium levels measured with colorimetric method and expressed in mg/dL.
Concentration of hydroperoxides serum levels (UCARR) | baseline
  The concentration of hydroperoxides serum levels is measured with dROMs test, a colorimetric method and expressed in UCARR. In the dROMs test the free radicals, primarily hydroperoxides, contained in the biological sample, close to iron, generate alkoxyl and peroxyl radicals, according to the Fenton's reaction. The radicals, reacting with a chromogenic mixture, oxidize it and transform it into a photo-metrically measurable coloured derivative. The values are expressed in arbitrary units (UCARR), 1 UCARR corresponding to 0.08 mg/100 mL of hydrogen peroxide.
Concentration of total antioxidant serum levels (µmol/L) | baseline
  The concentration of total antioxidant serum levels is measured with BAP-Test (Biological Antioxidant Potential). It measures the amount of endogenous and exogenous substances in plasma that have the potential to be antioxidants and can counteract radical species and is reported in µmol/L. In the BAP test, the biological antioxidant potential of plasma barrier is based on the ability of all antioxidants active to re-duce a colored solution of ferric ions (Fe3+) to ferrous ions (Fe2+), resulting a decoloration of the solution that is detectable photometrically
Measurement of Oxidative stress Index (dimensionless ratio) | baseline
  the Oxidative stress Index (OSI index), is a ratio calculated from BAP and dROMs (BAP/dROMs). The antioxidative/oxidative stress ratio was also calculated using the ratio equation: BAP/d-ROMs. According to literature, we named this ratio the OSI index, which is an index of potential antioxidant capacity. The criterion value for the BAP/d-ROMs ratio was set at 7.3. Accordingly, a value lower than 7.3 was defined as an oxidized type and a higher or equal one as a reduced type.
Nutritional Risk Index NRI | baseline
  The Nutritional Risk Index (NRI) is a tool designed to assess a patient's nutritional status and predict the risk of complications associated with malnutrition. It is calculated using the following formula:
  NRI = (1.519 × serum albumin [g/L]) + (41.7 × current weight [kg] / usual weight [kg]) The lower the score, the higher the risk. (No risk: NRI > 100- Severe risk: NRI < 83.5 )
Prognostic Nutritional Index (PNI) | baseline
  The Prognostic Nutritional Index (PNI) is a tool used to assess the immunological and nutritional status of patients, particularly in predicting surgical outcomes, cancer prognosis, and postoperative complications.The PNI is calculated using the following formula:
  PNI=(10×serum albumin (g/dL))+(0.005×total lymphocyte count per mm^3) The lower the score, the higher the risk.(Normal nutritional status, low risk: PNI > 38; moderate risk: scores between 35 and 38 severe malnutrition, high risk: PNI < 35).
Self-reported nutritional, psychological, and lifestyle survey | baseline
  Participants will complete an online survey including questions on general information, prevalence of medication, supplement, and nutraceutical use, body mass index (BMI), dietary habits, adherence to the Mediterranean diet, eating behavior, symptoms of malnutrition, psychological stress level, physical activity, and musculoskeletal disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Irene G Aprile, MD, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi, Centro Santa Maria della Provvidenza, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Di Vincenzo O, Marra M, Sammarco R, Speranza E, Cioffi I, Scalfi L. Body composition, segmental bioimpedance phase angle and muscular strength in professional volleyball players compared to a control group. J Sports Med Phys Fitness. 2020 Jun;60(6):870-874. doi: 10.23736/S0022-4707.20.10548-6. PMID 32487981
- [Background] Maggiora A, Lozeron H. [The role of the irradiation time in dermatological radiotherapy]. Dermatologica. 1966;133(1):21-7. No abstract available. French. PMID 5927356
- [Background] Campa F, Silva AM, Matias CN, Monteiro CP, Paoli A, Nunes JP, Talluri J, Lukaski H, Toselli S. Body Water Content and Morphological Characteristics Modify Bioimpedance Vector Patterns in Volleyball, Soccer, and Rugby Players. Int J Environ Res Public Health. 2020 Sep 10;17(18):6604. doi: 10.3390/ijerph17186604. PMID 32927903
- [Background] Sies H. Oxidative stress: a concept in redox biology and medicine. Redox Biol. 2015;4:180-3. doi: 10.1016/j.redox.2015.01.002. Epub 2015 Jan 3. PMID 25588755
- [Background] Vassalle C, Vigna L, Bianchi S, Maffei S, Novembrino C, De Giuseppe R, de Liso F, Vannucci A, Tirelli S, Maiavacca R, Bamonti F. A biomarker of oxidative stress as a nontraditional risk factor in obese subjects. Biomark Med. 2013 Aug;7(4):633-9. doi: 10.2217/bmm.13.49. PMID 23905900
- [Background] Silva AM. Structural and functional body components in athletic health and performance phenotypes. Eur J Clin Nutr. 2019 Feb;73(2):215-224. doi: 10.1038/s41430-018-0321-9. Epub 2018 Oct 4. PMID 30287933
- [Derived] Siotto M, Cocco C, Bertoncini C, Guerrini A, Habib V, Antonacci E, Ruco E, Aprile IG. One Health Approach to Nutritional Status and Well-Being in Food Supply Chain Workers: A Study Protocol. Int J Environ Res Public Health. 2026 Jan 11;23(1):99. doi: 10.3390/ijerph23010099. PMID 41595893